CLINICAL TRIAL: NCT00215436
Title: A 12-week Double-Blind, Parallel-Group, Placebo- and Active- Controlled Trial to Evaluate the Efficacy and Safety of Formoterol Fumarate Inhalation Solution 20 Mcg in the Treatment of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Trial to Evaluate the Efficacy and Safety of Formoterol Fumarate in the Treatment of Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director Clinical Affairs, Dey L.P.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201-065
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2008-04

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD; formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the investigational drug in comparison with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of COPD
* Current or prior history of cigarette smoking

Exclusion Criteria:

* Medical diagnosis of asthma
* Chest X-ray diagnostic of significant disease other than COPD
* Significant condition or disease other than COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345
Dates: Start 2005-03; Primary Completion 2005-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Measure of lung function

SECONDARY OUTCOMES:
Change in lung function, as well as vital signs
Physical Exam results, Adverse event reporting, etc

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Research Site, Jasper, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tuscon, Arizona
  - Research Site, Buena Park, California
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Stockton, California
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Tampa, Florida
  - Research Site, Woodstock, Georgia
  - Research Site, Hines, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Florence, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Henderson, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Camillus, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Cranston, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Nelson HS, Gross NJ, Levine B, Kerwin EM, Rinehart M, Denis-Mize K; Formoterol Study Group. Cardiac safety profile of nebulized formoterol in adults with COPD: a 12-week, multicenter, randomized, double- blind, double-dummy, placebo- and active-controlled trial. Clin Ther. 2007 Oct;29(10):2167-78. doi: 10.1016/j.clinthera.2007.10.007. PMID 18042473
- [Result] Gross NJ, Nelson HS, Lapidus RJ, Dunn L, Lynn L, Rinehart M, Denis-Mize K; Formoterol Study Group. Efficacy and safety of formoterol fumarate delivered by nebulization to COPD patients. Respir Med. 2008 Feb;102(2):189-97. doi: 10.1016/j.rmed.2007.10.007. PMID 18363201